CLINICAL TRIAL: NCT06169553
Title: The IRIS Program: A Novel Pathway to Optimize Treatment of Injection-related Infections for People Who Inject Drugs in Hamilton, Ontario
Brief Title: The Injection-Related InfectionS (IRIS) Program
Acronym: IRIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: HAMSMaRT (Unknown); Keeping Six (Unknown); YWCA Hamilton (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAH-23-012
Record Dates: First submitted 2023-11-23; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Peer Support; Injection-related Infections; Infections; People Who Infect Drugs (PWID)
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants in the IRIS program will be offered a one-stop, low-barrier combined care model to address their injection-related infections. Specific program components include: (1) Diagnosis and treatment of injection-related infections; (2) Substance use treatment (3) Peer support; and (4) Care coordination/systems navigation.
  Interventions: Other: Holistic injection-related injection treatment

INTERVENTIONS:
Other: Holistic injection-related injection treatment — Participants in the intervention group will be provided additional supports to address their social and medical needs, including infectious disease management, addictions medicine, peer support, and systems navigation. Each participant will receive individualized care depending on their unique needs.

SUMMARY:
People who inject drugs are at risk of injection-related infections, like abscesses or infective endocarditis. The Injection-Related InfectionS (IRIS) program hopes to improve treatment for participants by providing a low-barrier, one-stop shop model for people who inject drugs who experience injection-related infections to access more holistic and compassionate care. IRIS is a non-randomized clinical trial, meaning that it offers a specific program to eligible patients. This program offers care for substance use and infectious disease with additional peer support and systems navigation, if interested. The investigators anticipate enrolling 80 participants in the intervention and will follow participants throughout the infection treatment period (estimated 6-12 weeks). The investigators will collect information at the time of enrolment, at the 6-month mark, and monthly via electronic medical chart review. The investigators will use an interrupted time series analysis to evaluate the impact of the intervention on rates of treatment completion, emergency department visits, hospitalizations, and death, before versus after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or older
* Able to provide informed consent
* Presenting with a confirmed or suspected injection-related infection (including skin and soft tissue infections, osteomyelitis, infective endocarditis, Hepatitis C, HIV, etc)
* History of injection drug use within 3 months of recruitment
* Lives in Hamilton, Ontario

Exclusion Criteria:

-

Ages: 16 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of emergency department visits and hospital readmission | Within 30 days of initial hospital admission or program enrolment

SECONDARY OUTCOMES:
Completion of intended course of treatment for the injection-related infection | Within 6 months of initial hospital admission or program enrolment
  Investigators will record whether or not participants have completed the intended course of treatment for their injection-related infection (e.g. completed course of antibiotics - YES or NO).
Number of hospital readmissions specifically for the infection that was the primary reason for program enrolment | Within 90-days of hospital discharge or program enrolment
Number of emergency department visits | Within 90-days of hospital discharge or program enrolment
Number of new initiations or record of continuation of substance use treatment | Within 90-days of hospital discharge or program enrolment
Mortality rates | Within 6-months of hospital discharge or program enrolment
Rates of program drop-out and reasons for discontinuation | Within 6-months of hospital discharge or program enrolment

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - HAMSMaRT Clinic, Hamilton, Ontario
  - David Braley Health Science Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Keeping Six - collaborative organization — https://keepingsix.org/about/